CLINICAL TRIAL: NCT07113288
Title: Inspire UAS High AHI/High BMI Post-Approval Study
Brief Title: Inspire UAS High Apnea Hypopnea Index (AHI)/High Body Mass Index (BMI) Post-Approval Study
Acronym: AHIBMI PAS
Status: Recruiting | Type: Observational
Sponsor: Inspire Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-005
Record Dates: First submitted 2025-05-07; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Obstructive Sleep Apnea (OSA)
Keywords: Obstructive Sleep Apnea; OSA; Inspire; AHI
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- High AHI: Following patients with 65<AHI≤100 events/hr after Inspire Implantation for a period of 5 years
  Interventions: Device: Inspire® UAS System
- High BMI: Following patients with 32<BMI≤40 kg/m2 after Inspire Implantation for a period of 5 years
  Interventions: Device: Inspire® UAS System

INTERVENTIONS:
Device: Inspire® UAS System — Participants will be implanted with a commercially available Inspire® UAS System. In addition, participants will receive a patient remote which is used to initiate therapy each night.

SUMMARY:
The purpose of this observational clinical study is to provide evaluation of long-term safety and effectiveness in a newly expanded patient population including patients with a higher AHI and a higher BMI.

DETAILED DESCRIPTION:
This post-approval study is a condition of FDA approval and will collect long-term safety and effectiveness data on an expanded population that includes patients with very severe obstructive sleep apnea (65<AHI≤100 events/hr), as well as those with a higher BMI (32<BMI≤40 kg/m2). Participants will be implanted with a commercially available Inspire UAS System. In addition, participants will receive a patient remote which is used to initiate therapy each night.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years of age;
2. Subject has a diagnosis of severe OSA (65 ≤ AHI ≤ 100) based on a recent sleep study (within 12 months) OR Subject has a diagnosis of moderate to severe OSA (15≤AHI≤100) AND a baseline Body Mass Index of 32<BMI≤40 kg/m2;
3. Subject has documented failure of, or intolerance to, positive airway pressure treatments (such as CPAP or BPAP machines; NOTE: PAP failure is defined as an inability to eliminate OSA (AHI > 15 despite PAP usage). PAP intolerance is defined as the inability to use PAP (> 5 nights per week, 4 hours of usage per night) or unwillingness to use PAP (e.g. patient returns the PAP system after attempting to use it).
4. Subject is willing and able to have stimulation hardware permanently implanted and to use the patient remote to activate the stimulation;
5. Subject is willing and able to return for follow-up visits, undergo sleep studies (including in-lab and at-home), and complete questionnaires related to the study;
6. Subject is willing and able to provide informed consent.

Exclusion Criteria:

1. Subject has a combination of central + mixed apneas > 25% of the total apnea-hypopnea index (AHI) based on a recent sleep study (within 12 months);
2. Subject has any anatomical finding that would compromise the performance of upper airway stimulation, such as the presence of complete concentric collapse of the soft palate;
3. Subject has any condition or procedure that has compromised neurological control of the upper airway;
4. Subject is unable or does not have the necessary assistance to operate the patient remote;
5. Subject is pregnant or plans to become pregnant;
6. Subject has an implantable device that may be susceptible to unintended interaction with the Inspire System;
7. Subject has a terminal illness with life expectancy < 12 months;
8. Any other reason the investigator deems the subject is unfit for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A post-market sample selected from enrolling center's real-world patient population
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2032-01-01 (Estimated); Study Completion 2032-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Procedure and/or Device Related Adverse Events (Safety and Tolerability) | 5 years post-implant
  Procedure-related Adverse Events; Device-related Adverse Events

SECONDARY OUTCOMES:
Change in Apnea Hypopnea Index Over Time | 5 years post-implant
  Evaluation of improvement in Apnea Hypopnea Index (AHI) over time: baseline (pre-implant) AHI compared to AHI after implant (collected and reported at annual study visits)
Body Mass Index | 5 years post-implant
  Body Mass Index will be collected at each yearly follow-up visit.
Change in Oxygen Desaturation Index (ODI) Over Time | 5 years post-implant
  Evaluation of improvement in Oxygen Desaturation Index (ODI) over time: baseline (pre-implant) ODI compared to ODI after implant (collected and reported at annual study visits)
Change in T90 (defined as total sleep time spent with arterial oxygen saturation (SaO2) < 90%) Over Time | 5 years post-implant
  Evaluation of improvement in T90 (defined as total sleep time spent with arterial oxygen saturation (SaO2) < 90%) over time: baseline (pre-implant) T90 compared to T90 after implant (collected and reported at annual study visits)
Change in Epworth Sleepiness Scale (ESS) Over Time | 5 years post-implant
  Evaluation of improvement of Epworth Sleepiness Scale (ESS) over time: baseline (pre-implant) ESS compared to ESS after implant (collected and reported at annual study visits)

OTHER OUTCOMES:
Evaluation of Therapy Usage and Adherence Over Time | 5 years post-implant
  Therapy usage - reported as hours of use per week, is recorded by the Inspire UAS system and will be captured during the device check at the 6M and annual (1-5 year) study visits. This value will be used to quantify device use and adherence over time.
Change in Patient Satisfaction Over Time | 5 years post-implant
  A patient satisfaction survey, designed to collect information about the patient's experience with the Inspire UAS system, will be collected at the 6M and annual (1-5 year) study visits. This survey will provide information about relative satisfaction with the therapy over time.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Colorado ENT & Allergy, Colorado Springs, Colorado
  - Florida Sleep Specialists, Bradenton, Florida
  - Rush University Medical Center, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Rochester, Rochester, New York